CLINICAL TRIAL: NCT07081139
Title: Leveraging Deep Learning to Optimize the Individualized Application of Eye-tracking Devices for the Early-stage Visual Function Screening of Both Special Needs Children and Typical Preschoolers
Brief Title: Visual Function Screening System With Special Needs Children and Typical Preschoolers
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202403039RINA
Record Dates: First submitted 2025-06-17; First posted 2025-07-23 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-03

CONDITIONS: Visual Function; Vision; Special Needs Children
Keywords: Children; Ophthalmology
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General Population Group
  Interventions: Other: observational study, no interventional
- Special Needs Group
  Interventions: Other: observational study, no interventional

INTERVENTIONS:
Other: observational study, no interventional — no interventions

SUMMARY:
The early visual screening of children plays a critical role in promoting visual development, especially for those with visual impairments. Among various approaches, eye-tracking based visual assessment has emerged as a promising tool, particularly for infants, toddlers, and children with developmental disabilities who are unable to complete traditional vision tests. The object of this study is to design and investigate the effectiveness of using a deep learning based, individualized eye-tracking system to assess visual function, specifically visual acuity and visual field, in typical preschool children and infants under the age of three. This study aims to establish a reliable, noninvasive visual screening method that accommodates the diverse needs and abilities of young children.

DETAILED DESCRIPTION:
The investigators will recruit a total of 1,300 participants across four key groups to support the development and validation of an individualized visual function screening system using eye-tracking technology:

1. 300 adults to establish a reference dataset for gaze estimation models
2. 300 typically developing preschool children aged 3 to 5 years
3. 400 typically developing children under the age of 3
4. 300 children with special needs, including those with developmental disabilities and visual impairments Data collection will take place over 15 to 22 months, depending on the group.

ELIGIBILITY:
Inclusion Criteria:

* A. General Group 1. Inclusion Criteria

General adults:

1. Aged over 18 and under 70 years
2. Willing to undergo assessment and video recording using the "Deep Visual Tracking System"
3. Willing to sign the informed consent form

Typically developing preschool children aged 3 to 5:

1. Currently aged between 3 (inclusive) and 5 (inclusive) years
2. The primary caregiver agrees to allow the child to undergo assessment and video recording using the "Deep Visual Tracking System"

Children under 3 years old:

1. Currently under 3 years of age
2. The primary caregiver agrees to allow the child to undergo assessment and video recording using the "Deep Visual Tracking System"

2. Exclusion Criteria

General adults:

1. Presence of severe corneal disease or cataract that may interfere with data collection
2. Obvious abnormalities in eye or facial appearance, such as ptosis or facial trauma affecting facial structure

Typically developing preschool children aged 3 to 5:

1. Children with physical or mental disabilities
2. Children diagnosed with or suspected of having developmental delay
3. Children with obvious abnormalities in eye or facial appearance

Children under 3 years old:

(1) Children with physical or mental disabilities (2) Children diagnosed with or suspected of having developmental delay (3) Children with obvious abnormalities in eye or facial appearance

________________________________________ B. Special Needs Group

1. Inclusion Criteria (1) Children under the age of 12 with special needs, including physical, mental, or multiple disabilities (2) The primary caregiver agrees to allow the child to undergo assessment and video recording using the "Deep Visual Tracking System"
2. Exclusion Criteria (1) Children with refractive errors that are diagnosed by an ophthalmologist to significantly impair vision and are unable to wear corrective glasses during assessment (2) Children who are physiologically or emotionally unstable and unable to adapt and complete at least two assessment sessions

B. Special Needs Group

1. Inclusion Criteria (1) Children under the age of 12 with special needs, including physical, mental, or multiple disabilities (2) The primary caregiver agrees to allow the child to undergo assessment and video recording using the "Deep Visual Tracking System"

   Exclusion Criteria:
   * A. General Group
2. Exclusion Criteria

General adults:

1. Presence of severe corneal disease or cataract that may interfere with data collection
2. Obvious abnormalities in eye or facial appearance, such as ptosis or facial trauma affecting facial structure

Typically developing preschool children aged 3 to 5:

1. Children with physical or mental disabilities
2. Children diagnosed with or suspected of having developmental delay
3. Children with obvious abnormalities in eye or facial appearance

Children under 3 years old:

1. Children with physical or mental disabilities
2. Children diagnosed with or suspected of having developmental delay
3. Children with obvious abnormalities in eye or facial appearance

B. Special Needs Group 2. Exclusion Criteria

1. Children with refractive errors that are diagnosed by an ophthalmologist to significantly impair vision and are unable to wear corrective glasses during assessment
2. Children who are physiologically or emotionally unstable and unable to adapt and complete at least two assessment sessions

Ages: 0 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: General adults, typically developing preschool children aged 3 to 5 and under 3 years old. Additionally, children with special needs, regardless of the underlying cause, including those with physical or mental disabilities or multiple disabilities, such as autism spectrum disorder, cerebral palsy, visual impairments, and developmental delays.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Visual Acuity Classification by Deep Vision Tracking System (DVR System), Compared to Standard Clinical Assessment | 2 months
  Compare the DVR system's classification (normal vs. impaired vision) with results from standard clinical tests (e.g., Teller Acuity Cards). Report sensitivity and specificity. Cut-off values: logMAR 0.22 (Snellen decimal: 0.6) and 0.097 (Snellen decimal: 0.8).
Visual Field Detection Accuracy of the DVR System Compared to Standard Evaluation | 2 months
  This outcome assesses the accuracy of the DVR system in detecting visual field response in children, defined by whether the participant successfully fixates on screen-displayed peripheral stimuli. The DVR system's outputs will be compared to clinical observation. Accuracy will be evaluated via sensitivity and specificity.

SECONDARY OUTCOMES:
Criterion validity of DVR system visual acuity estimates (logMAR) | 2 months
  Compare DVR system logMAR estimates with clinical measurements (e.g., Teller Acuity Cards) using linear regression. Report slope coefficient; a slope near 1 indicates strong agreement. Target criterion: slope ≥ 0.8.
Test-retest reliability of DVR system visual acuity measurements | 2 months
  Participants will be re-tested within 2 weeks. Reliability will be assessed using standard error of measurement and coefficient of variation from panel data.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No